CLINICAL TRIAL: NCT02517827
Title: Percutaneous Intervention Versus Surgery in the Treatment of Common Femoral Artery Lesions A Prospective, Multi-centre, Randomised Study
Brief Title: Percutaneous Intervention Versus Surgery in the Treatment of Common Femoral Artery Lesions
Acronym: PESTO-AFC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Aljoscha Rastan, MD, Executive senior physician, Herz-Zentrums Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHZ_RASA_PESTO_1.0
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Artery Disease; Artery Stenosis
Keywords: common femoral artery; drug-coated balloon; surgical endarterectomy
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular procedure (Active Comparator): Common femoral artery (target lesion) to be treated with directional atherectomy and paclitaxel-coated balloon angioplasty. Optional: stentimplantation.
  Interventions: Device: Atherectomy and paclitaxel-coated balloon angioplasty
- Surgery (Active Comparator): Common femoral artery (target lesion) to be treated with open, surgical endarterectomy
  Interventions: Procedure: Open, surgical endarterectomy

INTERVENTIONS:
Device: Atherectomy and paclitaxel-coated balloon angioplasty — Directional atherectomy and paclitaxel-coated balloon angioplasty (optional with stentimplantation) of the common femoral artery
  Arms: Endovascular procedure
Procedure: Open, surgical endarterectomy — open, surgical endarterectomy of the common femoral artery
  Arms: Surgery

SUMMARY:
The endovascular therapy prevailed in nearly all regions of peripheral artery disease over open surgery techniques. However, in treatment of the common femoral artery vascular surgery is still the gold standard of therapy. One-year patency rates are between 90% and 95%. Today, only in selected cases an endovascular procedure for common femoral artery diseases is recommended.

The primary objective of this study is to compare the performance of directional atherectomy and drug-coated balloon angioplasty over vascular surgery in common femoral artery lesions in a prospective, multi-center, randomized clinical trial.

DETAILED DESCRIPTION:
Multicenter, prospective, randomized study to be conducted in centers in Europe. A total of 260 subjects will be entered into the study and will be randomized on a 1:1 basis to either directional atherectomy and drug coated balloon angioplasty (optional with stentimplantation), and surgical endarterectomy for treatment in symptomatic (Rutherford-Becker class 2 to 4) common femoral artery disease. All subjects will undergo repeat duplex-ultrasound measurements 6, 12, and 24 months to assess the primary endpoint of Binary Restenosis. Follow-up visits are scheduled 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be between 21 and 85 years old;
2. Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12-month angiographic evaluation;
3. Clinical diagnosis of symptomatic peripheral artery disease defined by Rutherford 2, 3, or 4;
4. Common femoral artery (CFA) stenosis (including CFA bifurcation) >70% (visual estimate) or occlusion; Additional non-target lesion(s) in remaining non-target vessel(s), except ipsilateral iliac arteries, can be treated at the physician´s discretion;
5. At least one vessel outflow (infrapopliteal arteries) to the foot (without stenosis >50%).
6. Endovascular Procedure: successful target lesion crossing of the guidewire (guidewire located intraluminally);
7. Non-target lesion interventions (TASC A and B) to restore adequate blood flow, in the same index procedure are allowed. This intervention must be prior to the treatment of the study lesion and successful;
8. Willing to comply with the specified follow-up evaluation;
9. Written informed consent prior to any study procedures.

Exclusion Criteria:

1. Ipsilateral significant (>50%) stenosis of the iliac arteries.
2. Significant (>50%) stenosis of all infrapopliteal arteries, no patent artery to the foot.
3. Angiographic evidence of thrombus within target vessel;
4. Thrombolysis within 72 hours prior to the index procedure;
5. In-Stent restenosis or restenosis of the native common femoral artery.
6. Aneurysm in the abdominal aorta or iliac arteries;
7. Concomitant hepatic insufficiency, thrombophlebitis, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy;
8. Recent MI or stroke < 30 days prior to the index procedure;
9. Life expectancy less than 24 months;
10. Known or suspected active infection at the time of the index procedure;
11. Known or suspected allergies or contraindications to aspirin, clopidogrel bisulfate (Plavix) and ticlopidine (Ticlid), heparin, or contrast agent;
12. Any significant medical condition which, in the investigator´s opinion, may interfere with the subject´s optimal participation in the study;
13. The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 month
  Primary patency of the common femoral artery defined as freedom from target lesion restenosis (luminal narrowing of ≥50%) detected with duplex-ultrasound. The definition of a 50% restenosis is based on the peak systolic velocity ratio >2.4.

SECONDARY OUTCOMES:
Primary patency | 24 month
  Primary patency of the common femoral artery defined as freedom from target lesion restenosis (luminal narrowing of ≥50%) detected with duplex-ultrasound. The definition of a 50% restenosis is based on the peak systolic velocity ratio >2.4.
target lesion revascularisation | 6, 12, and 24 month
  Need for target lesion revascularisation after index procedure

OTHER OUTCOMES:
Rutherford-Becker class | 6, 12, and 24 months
  Change in Rutherford-Becker class

CONTACTS AND LOCATIONS:
Overall Officials: Aljoscha Rastan, MD, Principal Investigator — aljoscha.rastan@universitaets-herzzentrum.de
Locations (1):
- Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Germany

REFERENCES:
- [Derived] Rastan A, Bohme T, Zeller T. Percutaneous intervention versus surgery in the treatment of common femoral artery lesions: study protocol for the prospective, multi-center, randomized PESTO-CFA trial. Trials. 2024 Jun 8;25(1):370. doi: 10.1186/s13063-024-08219-1. PMID 38851710